CLINICAL TRIAL: NCT01191073
Title: A Study on the Fit and Behaviour of Computer-aided Design and Rapid Prototyping Fabrication of Removable Partial Dentures
Brief Title: Manually Versus Digitally Fabricated Removable Partial Dentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009/655
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Partially Edentulous Patients
Keywords: edentulous
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAD/CAM fabricated dentures (Experimental): group receiving Computer-Aided Design/Computer-Aided Manufacturing (CAD/CAM)fabricated removable partial dentures (double blind)
  Interventions: Device: CAD/CAM fabricated RPD's
- traditional fabricated dentures (Active Comparator): group receiving traditional fabricated dentures (double blind)
  Interventions: Device: traditional fabricated RPD's

INTERVENTIONS:
Device: CAD/CAM fabricated RPD's — group receiving Computer-Aided Design/Computer-Aided Manufacturing (CAD/CAM)fabricated removable partial dentures (double blind)
  Arms: CAD/CAM fabricated dentures
Device: traditional fabricated RPD's — group receiving traditional fabricated dentures (double blind)
  Arms: traditional fabricated dentures

SUMMARY:
In the clinical trial, the Computer Aided Design/Computer Aided Manufacturing (CAD/CAM) fabricated removable partial dentures (RPD's) are evaluated on casts and clinically compared with a traditional fabricated RPD for 50 consecutive patients.

During 5 years the patients are in a follow-up program in order to judge long-term stability, loss of retention, fractures, … of both groups of dentures.

DETAILED DESCRIPTION:
The classic removable partial denture (RPD) is a denture fabricated in CrCo using the "lost wax" technique. This hand-made way of working makes the final result vulnerable, not always predictable and not reproducible.

Computer Aided Design/Computer Aided Manufacturing (CAD/CAM) techniques have been introduced in dentistry, particularly to fabricate crowns and bridges (fixed partial dentures). There is little research in the field of removable partial framework fabrication. This may be in part be attributed to the lack of suitable dedicated software.

In the technical part of the study, existing software and hardware is adjusted to maximize the automation in the application of computer-aided technologies to surveying of digital casts and pattern design and the subsequent production of sacrificial patterns using removable partial (RP) technologies.

In the clinical trial the CAD/CAM fabricated RPD's are evaluated on casts and clinically and compared with a traditional fabricated RPD for 50 consecutive patients. For every patient, two RPDs are made in the same material (CrCo).The clinical parameters (fit, stability, retention, support, friction) are double blind evaluated by two dentists. At the end of the treatment, the patient can choose one of them.

Both RPDs are fabricated in the same time frame for the fabrication of the "classic" RPD. There are for the patient no extra sessions scheduled.

During 5 years the patients are in a follow-up program in order to judge long-term stability, loss of retention, fractures, … of both groups of dentures.

Hypothesis1: CAD/CAM fabricated RPD's can meet the clinical standards for RPD's.

Hypothesis 2: Dentists do not observe a difference between the classic and CAD/CAM fabricated RPD.

Hypothesis 3: Patients do not see/feel any difference between the classic and CAD/CAM fabricated RPD.

ELIGIBILITY:
Inclusion Criteria:

* patients in need of a classic removable partial denture (RPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
fit of framework | 9 months
  After casting "fit of the framework" between two identical reomvable partial dentures (same design, looks, material...) fabricated in a different way.

SECONDARY OUTCOMES:
placement of RPD + control of placement | 3 to 5 days
  There will be a placement of a removable partial denture, and after 3 to 5 days, this placement will be re-checked as a follow up.
re-evaluation of the RPD placement | every 6 months, for 5 years
  Every 6 months, for 5 years, the RPD placement will be followed up.

CONTACTS AND LOCATIONS:
Overall Officials: Lieve Van Zeghbroeck, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium